CLINICAL TRIAL: NCT07172048
Title: Correlation Between Foot Pressure Distribution and Curve Pattern in Adolescent Idiopathic Scoliosis
Brief Title: This Cross-sectional Study Investigates the Relationship Between Different Curve Patterns in Adolescent Idiopathic Scoliosis (AIS) and the Distribution of Foot Pressure. It Aims to Determine Whether Coronal and Sagittal Curve Patterns Are Associated With Asymmetries in Plantar Pressure Distribution
Status: Active, not recruiting | Type: Observational
Sponsor: Mahmoud Ibrahim Elsayed Aly Mahmoud (Other)
Collaborators: Advanced Rehabilitation Center, Egypt (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Ibrahim Elsayed Aly Mahmoud, Lecturer, Advanced Rehabilitation Center, Egypt
Organization: Advanced Rehabilitation Center, Egypt (Other)
Other Study IDs: P.T.REC/012/005853
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis Idiopathic
Keywords: Scoliosis; Foot Pressure; Scoliosis Curve Pattern
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major Thoracic: The cohort will consist of adolescents aged 10-18 years diagnosed with adolescent idiopathic scoliosis (AIS), with Cobb angles ranging from 10° to 45°, and no prior surgical intervention. Participants will be recruited from orthopedic scoliosis clinics such as ARC for Physiotherapy. The study will involve non-invasive assessments including baropodometric foot pressure analysis and radiographic evaluation of scoliosis curve patterns. No therapeutic intervention will be applied; the study is observational and cross-sectional in nature.
  Interventions: Diagnostic Test: Foot pressure Distribution test
- Major Lumbar: The cohort will consist of adolescents aged 10-18 years diagnosed with adolescent idiopathic scoliosis (AIS), with Cobb angles ranging from 10° to 45°, and no prior surgical intervention. Participants will be recruited from orthopedic scoliosis clinics such as ARC for Physiotherapy. The study will involve non-invasive assessments including baropodometric foot pressure analysis and radiographic evaluation of scoliosis curve patterns. No therapeutic intervention will be applied; the study is observational and cross-sectional in nature.
  Interventions: Diagnostic Test: Foot pressure Distribution test

INTERVENTIONS:
Diagnostic Test: Foot pressure Distribution test — This study is observational and does not involve any therapeutic or experimental intervention. Participants will be divided into two groups based on their scoliosis curve pattern:
  Group 1: Adolescents with a major thoracic curve. Group 2: Adolescents with a major lumbar curve.
  Each participant will undergo non-invasive assessments including:
  Baropodometric foot pressure analysis during static standing to evaluate pressure distribution in both coronal and sagittal planes.
  Radiographic evaluation to classify curve patterns using Cobb's angle, Central Sacral Vertical Line, and Plumb Line.

SUMMARY:
This cross-sectional study investigates the relationship between different curve patterns in Adolescent Idiopathic Scoliosis (AIS) and the distribution of foot pressure. It aims to determine whether coronal and sagittal curve patterns are associated with asymmetries in plantar pressure distribution during static standing.

DETAILED DESCRIPTION:
Study Objectives Primary Objective: To assess the correlation between curve pattern and foot pressure percentage in the coronal plane.

Secondary Objective: To assess the correlation between curve pattern and foot pressure percentage in the sagittal plane.

Study Design Type: Observational (Cross-sectional) Model: two Group Time Perspective: Cross-Sectional Statistical Analysis: Pearson correlation coefficient will be used to determine the strength and direction of the relationship.

ELIGIBILITY:
Inclusion Criteria:

* • 1- Adolescents aged 10-18 years.

  * 2- Diagnosed with idiopathic scoliosis.
  * 3- Cobb angle between 10° and 45°.
  * 4- No prior surgical intervention for scoliosis.

Exclusion Criteria:

* • 1- Presence of congenital or neuromuscular scoliosis.

  * 2- Previous spinal surgery.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of adolescents aged 10 to 18 years diagnosed with adolescent idiopathic scoliosis (AIS). Participants will be divided into two groups based on their curve pattern:
  Group 1: Individuals with a major thoracic curve. Group 2: Individuals with a major lumbar curve.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Foot pressure distribution in adolescents with idiopathic scoliosis | 1-2 days
  measured using baropodometry during static standing.

SECONDARY OUTCOMES:
Correlation between curve pattern characteristics (e.g., Cobb angle, Central Sacral Vertical Line, Plumb Line) and foot pressure asymmetry. | 2 days
  Identification of any compensatory postural adaptations associated with different curve patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- ARC, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) collected during this study will be treated as confidential and will not be publicly shared. Data will be anonymized using unique participant codes to ensure privacy. Access to IPD will be restricted to the research team and authorized personnel involved in data analysis.
  No IPD will be shared with third parties or published in a way that could identify participants. Any future data sharing will require additional ethical approval and participant consent.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting documents (Study Protocol, SAP, ICF, CSR, Analytic Code) will be available starting January 2026, after initial data analysis is completed. They will remain accessible for 5 years, until December 2030, for academic and collaborative purposes upon request.
Access Criteria: Access to supporting information will be granted to academic researchers, clinicians, and collaborators with a legitimate interest in adolescent idiopathic scoliosis research. Requests must be submitted to the principal investigator and will be reviewed by the research team and ethics committee. Approved documents will be shared via secure institutional email or repository, ensuring confidentiality and ethical compliance.

REFERENCES:
- See also: This study showed that regional plantar foot pressure was significantly higher in AIS patients during quiet standing compared to healthy individuals. AIS patients also had increased pelvic height and altered center-of-pressure trajectories, suggesting po — https://link.springer.com/content/pdf/10.1007/s13530-014-0197-6.pdf